CLINICAL TRIAL: NCT04564222
Title: Double-Blind Cluster Randomized Controlled Trial of Chicken Liver and Eggshell Crackers in Mothers During Pregnancy and Lactation in a Disadvantaged Setting in Indonesia
Brief Title: Sustainable Intervention of Supplementation to Improve Kid's Growth Study
Acronym: SISTIK-G
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Collaborators: Universitas Padjadjaran (Other); University of Otago (Other); USDA, Western Human Nutrition Research Center (U.S. Federal Agency); VitMin Lab (Unknown); International Food Policy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 216447/Z/19/Z
Record Dates: First submitted 2020-09-20; First posted 2020-09-25 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Birth Length; Linear Growth; Micronutrients; Dietary Intakes
Keywords: Chicken Liver; Eggshell; Crackers; Pregnancy; Lactating Mother; Indonesia

STUDY DESIGN:
Intervention Model Description: A total of 324 pregnant women will be recruited from 28 clusters (villages) and will be randomised to either intervention or control using a randomized sequence, stratified by villages with < 100 and ≥ 100 infants using block sizes of 2 and 4. Selected pregnant women from these villages will receive daily interventions in the form of 75 gram food products, made from chicken liver and chicken eggshells (Micronutrient-enriched Crackers/MEC) or placebo. The MEC and placebo will be given from 8-14 weeks gestation to 5 months' post-partum.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micronutrient Enriched Crackers (MECs) (Experimental): Micronutrient Enriched Crackers (MECs) are a deep-fried snack product rich in iron, zinc, calcium, and vitamin A made from chicken liver and chicken eggshell powder.
  Consume daily, 75 gram/day, during pregnancy (from 8-14 weeks gestation to delivery) and lactation (from delivery to 5 months post-partum).
  Interventions: Dietary Supplement: Micronutrient Enriched Crackers (MECs)
- Placebo (Placebo Comparator): Placebo Crackers are a deep-fried snack product made from the basic cracker ingredients (mainly wheat flour) with the addition of Pangium edule seeds to provide a color similar to the intervention product (MECs).
  Consume daily, 75 gram/day, during pregnancy (from 8-14 weeks gestation to delivery) and lactation (from delivery to 5 months post-partum).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Micronutrient Enriched Crackers (MECs) — MECs are manufactured according to the Standard Operational Procedures which have been developed taking into account the Hazard Analysis and Critical Control Point (HACCP) to maintain quality and safety and ensure the "Ready-to-eat MEC products" are safe. Data on the micronutrient concentrations and any potential bacteriological (Salmonella sp is negative, Bacillus cereus, Enterobacteriaceae, and Coagulase positive streptococci level are considered safe) and chemical contaminants (Pb, Hg, Cd, As, and Sn are not detectable) in the MEC products have been obtained from analysis in the laboratory of Saraswanti Indo Genetech, which has been accredited by KAN LP-184-IDN with SNI ISO/IEC 17025: 2008. Laboratory analysis of MEC products will be repeated at the middle and the end of the RCT to check on the quality and safety of the MEC product.
  Other Names: SISTIK
  Arms: Micronutrient Enriched Crackers (MECs)
Dietary Supplement: Placebo — Placebo crackers are manufactured according to SOPs which have been developed taking into account the HACCP to maintain quality and safety and ensure the "Ready-to-eat placebo products" are safe. Data on the micronutrient concentrations and any potential bacteriological (Salmonella sp is negative, Bacillus cereus, Enterobacteriaceae, and Coagulase positive streptococci level are considered safe) and chemical contaminants (Pb, Hg, Cd, As, and Sn are not detected) in the placebo have been obtained based on the analysis in the laboratory of Saraswanti Indo Genetech, which has been accredited by KAN LP-184-IDN with SNI ISO/IEC 17025: 2008. Laboratory analysis of placebo samples will be repeated at the middle and the end of the RCT to check on the quality and safety of the placebo product.
  Arms: Placebo

SUMMARY:
Our earlier research has highlighted a high prevalence of anaemia, micronutrient deficiencies, and impaired infant growth among lactating women and infants in Sumedang district, West Java, Indonesia that were associated with large deficits in their micronutrient intakes. In response to these disturbing findings we have developed the micronutrient- enriched crackers (MEC) based on powdered eggshells and chicken liver, a readily available and affordable, local animal-source food. We will supply these MEC or a placebo, manufactured locally, weekly to a group of women in Sumedang district from 8-14 weeks gestation to 5 months post-partum in an effort to enrich the micronutrient content of the daily diets of the treatment group so they no longer have any dietary shortfalls in micronutrients. Our overall aim is to determine if MEC consumed daily by mothers for 6 months during pregnancy improves the birth length of their infants, and if daily consumption of MEC is continued daily to 5 months post-partum enhances infant linear growth compared to the placebo.

This study is funded by the UK Wellcome Trust, the grant reference number is 216447/Z/19/Z.

DETAILED DESCRIPTION:
A double-blind two-phase cluster randomized controlled trial (RCT) will be conducted in West Java, Indonesia to determine whether daily consumption of MEC from 8-14 weeks' gestation to delivery improves birth length compared to placebo (Phase 1) and whether daily consumption of MEC from 8-14 weeks gestation to 5 months post-partum improves attained linear growth of infants at age 5 months and linear growth velocity of infants from birth to age 5 months compared to placebo (Phase 2). A total of 324 pregnant women will be recruited through midwives/public health centre from 28 clusters (villages) in Sumedang district. Clusters will be randomly assigned to receive placebo or micronutrient- enriched crackers (MEC) daily, distributed by cadres from 8-14 weeks gestation to 5 months post-partum. Women who fulfil trial criteria will be invited to participate in the RCT.

Placebo and MEC (based on powdered eggshells and chicken liver) will be manufactured locally according to Standard Operational Procedures (SOPs), so they are identical in size, color, and packaging, with a code known only by the local production manager. The code will not be shared until the primary outcome has been analysed statistically or if requested by the Ethics Committee and/or Data Safety Monitoring Board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Gestational age 7-13 weeks at the time of the screening process and be willing to take part in an intervention study at 8-14 weeks gestation
* Permanent residents who do not plan to move in the next 1 year

Exclusion Criteria:

* Mothers who have chronic diseases such as hypertension (blood pressure > 140/90 mmHg) or under treatment for hypertension, diabetes (non-fasting blood sugar > 200 mg/dL)/ under treatment for diabetes, hypercholesterolemia (blood total cholesterol > 240 mg/dL), hyperuricemia (blood uric acid > 6 mg/dL), have had a history of tuberculosis or under treatment for tuberculosis; or under treatment for other chronic diseases that required a long treatment, such as cancer, heart disease, epilepsy, etc.
* Have a history of preeclampsia/eclampsia and gestational diabetes in their previous pregnancy
* Have a risk of chronic energy deficiency (mid-upper arm circumference < 23.5 cm)
* Have severe anaemia (haemoglobin < 70 g/L or < 7 g/dL)
* Have a history of allergy to chicken liver and/or eggs

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Birth length | 24 hours after birth
  All measurements will be taken to the nearest millimetre (mm) using standardized techniques and trained anthropometrists using a portable infantometer (SECA 417, measuring range: 10-100 cm). The measurements will be made on nude infants and will be recorded in duplicate, or triplicate if the difference between the first and second measurement is more than the recommended range (i.e., 7 mm).
Attained linear growth and growth velocity | 5 months (+/- 1 week) post partum
  All length measurement will be taken to the nearest millimetre (mm) using standardized techniques by trained anthropometrists using a portable infantometer (SECA 417, measuring range: 10-100 cm) The measurements will be made on nude infants and will be recorded in duplicate, or triplicate if the difference between the first and second measurement is more than the recommended range (i.e., 7 mm).

SECONDARY OUTCOMES:
Birth weight | 24 hours after birth
  All weight measurements will be taken to the nearest 10 grams using standardized protocols by trained anthropometrists using an electronic scale (SECA 334). The measurements will be made on nude infants and will be recorded in duplicate, or triplicate if the difference between the first and second measurement is more than the recommended range (i.e., 100g).
Maternal haemoglobin level | 35-36 gestational age and 5 months (+/- 1 week) post partum
  Blood will be taken by a trained personnel and hemoglobin concentration (g/dL) in the mother will be analysed by complete blood count in a certified laboratory (Prodia Laboratory; Sysmex XN-1000).
Maternal food intake | 35-36 weeks gestational age, 2 months (+/- 1 week) and 5 months (+/- 1 week) post partum
  Weighed records will be collected by the mothers on 3 non-consecutive days: 2 weekdays and 1 weekend day using a digital scale with precision of 4 grams (Kitchen Scale EK3131). On the next day after each weighed food record has been completed by the mother, an experienced research assistant will conduct a 24-hour recall on the mother using telephone/online communication. Results from the weighed record and recall will be combined to determine maternal food intake, which will be converted into nutrient intakes based on the weight and nutritional value of each food using the Indonesian Food Composition Table. The Multiple Source Method (MSM) program will be applied to estimate individual usual intakes of energy and nutrients as well as the usual intake distributions for the study population.
Status of breastfed infants (exclusive vs. non-exclusive) and breast milk volume | 5 months (+/- 1 week) post partum
  The deuterium dose-to-the mother technique will be performed to measure the volume of breast milk consumed by the infants and the status of breastfed infants. As much as 30 grams of Deuterium Oxide (D2O) are taken by the mother orally, which is then excreted into the breast milk consumed by the infant. Saliva sampling will be carried out according to protocol guidelines established by the International Atomic Energy Agency (IAEA; Human Health Series No. 7) with some adjustments to the number of days of sampling. Maternal and infant saliva samples will be taken on the 0th day before the mother is given D2O dose, and subsequently post-dose on day 2 or 3, day 8 or 9, and on day 13 or 14. A total of 2 mL of maternal and 1 mL of infant saliva will be collected on each sampling day. Saliva will be analyzed using Fourier Transform Infrared Spectrometry (FTIR), from which exclusive breastfeeding categorization and breast milk volume will be calculated using the Microsoft Excel Spreadsheet.
Breast milk micronutrient concentration | 5 months (+/- 1 week) post partum
  Full breast milk samples will be collected by mothers from one breast (washed with distilled, deionised water) using acid washed breast milk pumps (Medela Harmony Manual Breast Pump) into acid washed glass bottles. Mothers will be requested to refrain from breastfeeding on one breast at least 2 hours before the scheduled breast milk collection to allow for the collection of fore- and hindmilk.
  Breast milk micronutrient concentrations, including Na, Mg, P, K, Ca, Fe, Cu, Zn, Se will be analysed using ICP- MS Agilent 7900; Free Thiamine, TMP, and TPP using HPLC-FLD Agilent 1200; Cobalamin using Competitive Chemiluminescent Enzyme Immunase IMMULITE 1000; Riboflavin, FAD, FMN, NAD, panthothenic acid, pyridoxal, pyridoxine, biotin using UPLC-MS with a Waters ACQUITY UPLC I-Class system coupled to a Sciex 4500 triple quadrupole mass spectrometer; Performed retinol, Alpha-carotene, Beta-carotene, Beta-cryptoxanthin, Alpha- tocopherol, and Gamma-tocopherol using HPLC Agilent 1260.
Infant breast milk micronutrient intake | 5 months (+/- 1 week) post partum
  Data generated from the volume of infant's breast milk intake using Deuterium Oxide Dose-to- Mother Technique and analyzed breast milk micronutrient concentrations will be used to calculate breast milk micronutrient intakes of the infants at 5 months post-partum.
Maternal micronutrient status | 35-36 weeks gestational age and 5 months (+/- 1 week) post partum
  Data generated from maternal micronutrient concentrations in serum (Ferritin, Soluble Transferrin Receptor (sTfR), Retinol-Binding Protein (RBP), Zn, and Se) and adjusted for inflammation status, where appropriate, using C-reactive protein and Alpha-1-acid glycoprotein will be used to assess maternal micronutrient status.
  The cutoffs used to define deficiency for each maternal biomarker will be as follows: adjusted serum ferritin, < 15 μg/L; adjusted sTfR, > 8.3 mg/L; adjusted zinc < 10.7 μmol/L; adjusted RBP < 1.20 μmol/L; and adjusted selenium < 0.82 μmol/L.
Infant micronutrient status | 5 months (+/- 1 week) post partum
  Data generated from infant's serum micronutrient concentrations (Ferritin, sTfR, RBP, Zn, and Se) at 5 months post- partum, adjusted for inflammation status, where appropriate using C-reactive protein and Alpha-1-acid glycoprotein will be used to assess infant micronutrient status at 5 months post-partum.
  The cutoffs used to define deficiency for each biomarker among the infants will be as follows: adjusted ferritin, < 12 μg/ L, adjusted sTfR, > 8.3 mg/L; adjusted zinc < 9.9 μmol/L; adjusted RBP < 0.83 μmol/L (27); adjusted selenium < 0.82 μmol/L; vitamin B12 < 148 pmol/L.
Morbidity incidence rate of mothers and infant | 14 weeks and 31-32 weeks gestational age, 1 month (+/- 1 week) and 4 months (+/- 1 week) post partum
  The morbidity calendar for both mother and infant will be recorded by respondents independently and checked by research cadres once a week. The maternal morbidity calendar will be recorded over one month (for seizure, fever, headache, diarrhea, vaginal bleeding, cough, sore throat) at 14 weeks and 31-32 weeks of gestation, and 1 month and 4 months post-partum (for diarrhea, fever, cold, cough, vomit, ear infection, sore throat). The infant morbidity calendar will also be recorded over one month when the infant is 1 month and 4 months post-partum (for diarrhoea, fever, cold, cough, vomit, ear infection, sore throat). Digital thermometers will be provided to the respondents for self assessment of maternal and infant fever.

CONTACTS AND LOCATIONS:
Overall Officials: Aly Diana, PhD, Principal Investigator — SEAMEO Regional Centre for Food and Nutrition
Locations (1):
- Tanjungsari, Pamulihan, and Sukasari Subdistrict, Sumedang, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Birth length and birth weight to analyse factors associated with stunting, underweight, and wasting; exclusively breastfed infant status confirmed by deuterium oxide dose to mother technique; micronutrient status of the lactating mother and their infant; maternal dietary intake and prevalence of inadequate intakes during pregnancy and lactation; the volume of exclusively breastfed infants and non-compliers; micronutrient concentrations of breastmilk; the effectiveness of MEC during pregnancy and lactation.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after analysis has been finalised (around the end of February 2024) and available for a long term.
Access Criteria: Data will be shared through open journal repositories; free source data sharing (Open Science Framework); harmonised maternal dietary intake will be available to the Food and Agriculture Organization of the United Nations - Global Individual Food consumption data Tool (FAO/WHO GIFT) platform; shared data available in South East Asia Ministers of Education Organization Regional Centre for Food and Nutrition (SEAMEO RECFON) website and social media; use of MEC permitted for non-commercial purposes under a creative common license.

REFERENCES:
- [Background] Daniels L, Gibson RS, Diana A, Haszard JJ, Rahmannia S, Luftimas DE, Hampel D, Shahab-Ferdows S, Reid M, Melo L, Lamers Y, Allen LH, Houghton LA. Micronutrient intakes of lactating mothers and their association with breast milk concentrations and micronutrient adequacy of exclusively breastfed Indonesian infants. Am J Clin Nutr. 2019 Aug 1;110(2):391-400. doi: 10.1093/ajcn/nqz047. PMID 31152543
- [Background] Diana A, Haszard JJ, Purnamasari DM, Nurulazmi I, Luftimas DE, Rahmania S, Nugraha GI, Erhardt J, Gibson RS, Houghton L. Iron, zinc, vitamin A and selenium status in a cohort of Indonesian infants after adjusting for inflammation using several different approaches. Br J Nutr. 2017 Nov;118(10):830-839. doi: 10.1017/S0007114517002860. PMID 29189196
- [Background] Diana A, Mallard SR, Haszard JJ, Purnamasari DM, Nurulazmi I, Herliani PD, Nugraha GI, Gibson RS, Houghton L. Consumption of fortified infant foods reduces dietary diversity but has a positive effect on subsequent growth in infants from Sumedang district, Indonesia. PLoS One. 2017 Apr 20;12(4):e0175952. doi: 10.1371/journal.pone.0175952. eCollection 2017. PMID 28426828
- [Background] Domellof M, Dewey KG, Lonnerdal B, Cohen RJ, Hernell O. The diagnostic criteria for iron deficiency in infants should be reevaluated. J Nutr. 2002 Dec;132(12):3680-6. doi: 10.1093/jn/132.12.3680. PMID 12468607
- [Background] Dror DK, Allen LH. Overview of Nutrients in Human Milk. Adv Nutr. 2018 May 1;9(suppl_1):278S-294S. doi: 10.1093/advances/nmy022. PMID 29846526
- [Background] Dror DK, Allen LH. Retinol-to-Fat Ratio and Retinol Concentration in Human Milk Show Similar Time Trends and Associations with Maternal Factors at the Population Level: A Systematic Review and Meta-Analysis. Adv Nutr. 2018 May 1;9(suppl_1):332S-346S. doi: 10.1093/advances/nmy021. PMID 29846525
- [Background] Duizer LM, Diana A, Rathomi HS, Luftimas DE, Rahmannia S, Santi W, Nugraha GI, Haszard JJ, Gibson RS, Houghton LA. An Acceptability Trial of Desiccated Beef Liver and Meat Powder as Potential Fortifiers of Complementary Diets of Young Children in Indonesia. J Food Sci. 2017 Sep;82(9):2206-2212. doi: 10.1111/1750-3841.13807. Epub 2017 Jul 26. PMID 28746725
- [Background] Engle-Stone R, Haskell MJ, Ndjebayi AO, Nankap M, Erhardt JG, Gimou MM, Brown KH. Plasma retinol-binding protein predicts plasma retinol concentration in both infected and uninfected Cameroonian women and children. J Nutr. 2011 Dec;141(12):2233-41. doi: 10.3945/jn.111.145805. Epub 2011 Nov 2. PMID 22049292
- [Background] Gibson RS, Hotz C. Dietary diversification/modification strategies to enhance micronutrient content and bioavailability of diets in developing countries. Br J Nutr. 2001 May;85 Suppl 2:S159-66. doi: 10.1079/bjn2001309. PMID 11509105
- [Background] Human energy requirements: report of a joint FAO/ WHO/UNU Expert Consultation. Food Nutr Bull. 2005 Mar;26(1):166. No abstract available. PMID 15810802
- [Background] Institute of Medicine (US) Panel on Micronutrients. Dietary Reference Intakes for Vitamin A, Vitamin K, Arsenic, Boron, Chromium, Copper, Iodine, Iron, Manganese, Molybdenum, Nickel, Silicon, Vanadium, and Zinc. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222310/ PMID 25057538
- [Background] Institute of Medicine (US) Committee to Review Dietary Reference Intakes for Vitamin D and Calcium; Ross AC, Taylor CL, Yaktine AL, Del Valle HB, editors. Dietary Reference Intakes for Calcium and Vitamin D. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK56070/ PMID 21796828
- [Background] International Zinc Nutrition Consultative Group (IZiNCG); Brown KH, Rivera JA, Bhutta Z, Gibson RS, King JC, Lonnerdal B, Ruel MT, Sandtrom B, Wasantwisut E, Hotz C. International Zinc Nutrition Consultative Group (IZiNCG) technical document #1. Assessment of the risk of zinc deficiency in populations and options for its control. Food Nutr Bull. 2004 Mar;25(1 Suppl 2):S99-203. No abstract available. PMID 18046856
- [Background] Liu Z, Diana A, Slater C, Preston T, Gibson RS, Houghton L, Duffull SB. Development of a nonlinear hierarchical model to describe the disposition of deuterium in mother-infant pairs to assess exclusive breastfeeding practice. J Pharmacokinet Pharmacodyn. 2019 Feb;46(1):1-13. doi: 10.1007/s10928-018-9613-x. Epub 2018 Nov 14. PMID 30430351
- [Background] Liu Z, Diana A, Slater C, Preston T, Gibson RS, Houghton L, Duffull SB. Development of a Parsimonious Design for Optimal Classification of Exclusive Breastfeeding. CPT Pharmacometrics Syst Pharmacol. 2019 Aug;8(8):596-605. doi: 10.1002/psp4.12428. Epub 2019 Jul 3. PMID 31215140
- [Background] Michaelsen KF, Hoppe C, Roos N, Kaestel P, Stougaard M, Lauritzen L, Molgaard C, Girma T, Friis H. Choice of foods and ingredients for moderately malnourished children 6 months to 5 years of age. Food Nutr Bull. 2009 Sep;30(3 Suppl):S343-404. doi: 10.1177/15648265090303S303. PMID 19998864
- [Background] Rahmannia S, Diana A, Luftimas DE, Gurnida DA, Herawati DMD, Houghton LA, Gibson RS. Poor dietary diversity and low adequacy of micronutrient intakes among rural Indonesian lactating women from Sumedang district, West Java. PLoS One. 2019 Jul 11;14(7):e0219675. doi: 10.1371/journal.pone.0219675. eCollection 2019. PMID 31295313
- [Background] Schaafsma A, Pakan I, Hofstede GJ, Muskiet FA, Van Der Veer E, De Vries PJ. Mineral, amino acid, and hormonal composition of chicken eggshell powder and the evaluation of its use in human nutrition. Poult Sci. 2000 Dec;79(12):1833-8. doi: 10.1093/ps/79.12.1833. PMID 11194049
- [Background] Thomson CD. Assessment of requirements for selenium and adequacy of selenium status: a review. Eur J Clin Nutr. 2004 Mar;58(3):391-402. doi: 10.1038/sj.ejcn.1601800. PMID 14985676
- [Derived] Diana A, Rahmannia S, Suhadi YZ, Luftimas DE, Rizqi H, Purnamasari AD, Jihadillah A, Ansari MB, Haq DAZ, Pratiwi AN, Puspita DN, Affandy YIKD, Frampton CMA, Fahmida U, Houghton LA, Gibson RS. Chicken liver and eggshell crackers are a safe and affordable animal source food for overcoming micronutrient deficits during pregnancy and lactation in Indonesia: a double-blind, cluster randomized controlled trial (SISTIK Growth Study). BMC Pregnancy Childbirth. 2025 Aug 6;25(1):817. doi: 10.1186/s12884-025-07899-0. PMID 40770284
- [Derived] Zuhairini Y, Suryanto AH, Adnani QES, Anshari MB, Rizqi H, Fathonah A, Purnamasari AD, Pangasih AH, Jihadillah A, Puspita DN, Luftimas DE, Rahmannia S, Fahmida U, Gibson R, Diana A. Acceptability trial of local Indonesian snack (SISTIK) enriched with chicken liver and eggshell powder as a potential food to increase micronutrient intakes among women of reproductive age. Wellcome Open Res. 2025 Feb 24;9:550. doi: 10.12688/wellcomeopenres.20292.2. eCollection 2024. PMID 40093311
- [Derived] Diana A, Rahmannia S, Suhadi YZ, Luftimas DE, Rizqi H, Purnamasari AD, Jihadillah A, Ansari MB, Haq DAZ, Pratiwi AN, Scott S, Hampel D, Allen LH, Haszard JJ, Houghton LA, Gibson RS, Fahmida U. Chicken liver and eggshell crackers as a safe and affordable animal source food for overcoming micronutrient deficits during pregnancy and lactation in Indonesia: a double-blind, randomised placebo-controlled trial (SISTIK Growth Study). Wellcome Open Res. 2022 Jun 9;7:167. doi: 10.12688/wellcomeopenres.17879.1. eCollection 2022. PMID 35865219
- See also: International Atomic Energy Agency. Stable isotope technique to assess intake of human milk in breastfed infants. Human Health Series No. 7. Vienna: IAEA, 2010. — https://www-pub.iaea.org/MTCD/Publications/PDF/Pub1429_web.pdf
- See also: World Health Organization. Serum ferritin concentrations for the assessment of iron status and iron deficiency in populations. Vitamin and Mineral Nutrition Information System. Geneva: WHO, 2011 (WHO/NMH/NHD/MNM/112). — https://apps.who.int/iris/handle/10665/85843

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT04564222/SAP_000.pdf